CLINICAL TRIAL: NCT01101399
Title: Randomised Controlled Open-label Study to Evaluate Efficacy & Safety of Intravenous Ferric Carboxymaltose Versus no Treatment in Anaemic Subjects With Lymphoid Malignancies & Functional Iron Deficiency Receiving Chemotherapy
Brief Title: Ferric Carboxymaltose in Subjects With Functional Iron Deficiency Undergoing Chemotherapy
Acronym: FID-CHEMO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FER-FID-CHEMO
Record Dates: First submitted 2010-03-30; First posted 2010-04-09 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Iron-Deficiency Anemia
Keywords: Anemia; Lymphoproliferative Disorders; Chemotherapy; ferric carboxymaltose; iron
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia; Lymphoproliferative Disorders | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferric carboxymaltose (Active Comparator): Subjects will receive a total dose of 1,000 mg iron as FCM on the day of the next scheduled chemotherapy cycle after randomisation or continuous chemotherapy. In subjects with weight ≤66 kg, the first dose iron will be 500 mg; the second dose (500 mg) will be administered on the visit 4 (week 2).
  Interventions: Drug: Ferric carboxymaltose
- Local standard of care. (No Intervention): Subjects will be treated according to the local institutional practice.

INTERVENTIONS:
Drug: Ferric carboxymaltose — Subjects will receive a single dose of 1,000 mg iron as FCM infusion at baseline.
  Subjects of bw ≤66 kg will receive a single dose of 500 mg iron as FCM infusion at baseline (Week 0) and at Visit 4 (Week 2).
  Ferric carboxymaltose will be administered on the same day with chemotherapy treatment or within 24 hours before or after the chemotherapy. For subjects with bw ≤66 kg, if no chemotherapy planned for the visit 4 (Week 2), the second FCM dose should be infused independent of chemotherapy.
  Other Names: Ferinject
  Arms: Ferric carboxymaltose

SUMMARY:
Anaemia and functional iron deficiency are common conditions in patients with lymphoid malignancies, conditions which reduce significantly the quality of life and increase morbidity and mortality. Traditionally, Erythropoiesis Stimulating Agents (ESAs) have been used, but recently their use has been shown to have a negative impact on overall survival in different oncology populations. Recently published data suggest that intravenous (IV) iron can be effective in anaemia treatment, even without ESAs. This exploratory study is the first clinical project with ferric carboxymaltose (FCM) in patients with lymphoid malignancies: the data generated may be used for further evaluations of the drug in larger populations. In this study, 1,000 mg of IV iron as FCM will be administered on the same day or within 24 hours before or after chemotherapy treatment. The primary objective is to evaluate the efficacy of FCM in the correction of haemoglobin levels in anaemic subjects with lymphoid malignancies, undergoing chemotherapy. Secondary objectives aim to describe the safety and tolerability of FCM, and the effect of FCM treatment on iron status variables in subjects suffering from lymphoid malignancies.

DETAILED DESCRIPTION:
Multicentre, randomised, controlled, 2-arm open-label prospective pilot study to evaluate efficacy and safety of FCM in the treatment of anaemia in LPD subjects with functional iron deficiency (FID), undergoing chemotherapy. The subjects will be screened for eligibility within 4 weeks prior to inclusion to receive intravenous (IV) infusions of FCM or no FCM infusions (the subjects may be treated according to the local institutional practice if requiring symptomatic management of anaemia). After randomisation, the visits are scheduled weekly until Week 8.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (male or female) aged ≥18, suffering from indolent non-Hodgkin's lymphoma, multiple myeloma or chronic lymphocytic leukaemia on any chemotherapy excluding anthracycline containing.
* Life expectancy at least 6 months.
* Received at least 12 weeks (or 3 cycles) of treatment in the current course of chemotherapy before start of iron therapy.
* 8.5 g/dL Hb 10.5 g/dL at time of randomisation.
* Iron-restricted erythropoiesis as defined:

  * Stainable iron in bone marrow combined with transferrin saturation (TSAT) ≤20% OR
  * where the evaluation of stainable iron in bone marrow is not possible or available:

    * ferritin >30 ng/mL (women) or >40 ng/mL (men) and
    * TSAT ≤20%
* Signed informed consent (before any study procedure).
* Females of child-bearing potential must have a negative urine pregnancy test.

Exclusion Criteria:

* Any anaemia treatment within 4 weeks before inclusion (including red blood cell transfusion, ESA treatment and any oral/parenteral iron supplementation).
* Subjects weighing <35 kg.
* Subjects with increase in Hb during the chemotherapy (>1 g/dL rise between initiation of CT and screening laboratory value).
* Folate deficiency (serum folate <4.5 nmol/L) and/or vitamin B12 deficiency (serum cobalamin <145 pmol/L).
* Ongoing haemolysis defined as serum haptoglobin <0.2 g/L.
* Recent significant bleeding/surgery.
* Monotherapy with immunotherapy agents.
* Known chronic renal failure, creatinine >125 μmol/L.
* Anthracycline containing chemotherapy regimens.
* Clinically relevant active inflammatory disease other than the malignant disease (according to the judgement of the Investigator).
* Clinically relevant ongoing infectious disease including known human immunodeficiency virus.
* Serum-ferritin >800 ng/mL.
* Ongoing significant neurological or psychiatric disorders including psychotic disorders or dementia.
* Significant cardiovascular disease prior to study inclusion including myocardial infarction within 12 months prior to study inclusion, congestive heart failure New York Heart Association (NYHA) Grade III or IV, or poorly controlled hypertension according to the judgment of the Investigator.
* Elevation of liver enzymes (aspartate aminotransferase, alanine aminotransferase) over 3 times above the normal range or known acute hepatic disorder.
* Subject currently is enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study(ies), or subject is receiving other investigational agent(s).
* Females who are evidently pregnant (e.g., positive HCG test) or are breast feeding.
* Subject is not using adequate contraceptive precautions. Adequate contraceptive precautions are defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intra-uterine devices, sexual abstinence or vasectomised partner. Non-childbearing potential includes being surgically sterilised at least 6 months prior to the study or post menopausal, defined as amenorrhea for at least 12 months.
* Subject has known sensitivity to any of the products to be administered during dosing.
* Subject will not be available for follow-up assessment.
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-05; Primary Completion 2012-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in haemoglobin from baseline to Week 4 | Weeks 4 post baseline

SECONDARY OUTCOMES:
The percentage of subjects with blood haemoglobin increase of at least 1 g/dL in the absence of any red cell transfusion or ESA treatment. | 12 weeks post baseline
Change in haemoglobin from baseline to Week 6 | 6 weeks after baseline
Change in haemoglobin from baseline to Week 8 | 8 weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Torbjörn Karlsson, MD, PhD, Principal Investigator — Capio St Görans Sjukhus, Stockholm; Morgan McNamara, Study Director — Vifor Pharma, CH-8152 Glattbrugg, Switzerland
Locations (2):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany
- Department of Medicine, St Görans Hospital (Capio St Görans Sjukhus), Stockholm, Sweden